CLINICAL TRIAL: NCT04283552
Title: An Exploration of Gated and Non-Gated Dynamic PET/CT Imaging
Brief Title: Gated and Non-Gated Dynamic PET/CT Imaging
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Loss of funding
Sponsor: Washington University School of Medicine (Other)
Collaborators: Siemens Corporation, Corporate Technology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201910076
Record Dates: First submitted 2020-02-20; First posted 2020-02-25 (Actual); Results first posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Dynamic PET/CT Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Dynamic PET Imaging (Experimental): * Dynamic PET/CT imaging will begin at approximately the same time as the clinically prescribed radiotracer injection and will continue until approximately the start of the clinical scan
  * A subset of patients (up to 30 scheduled to undergo FDG or DOTATATE PET/CT imaging) will be asked to return within 7 days for a repeat imaging study.
  Interventions: Device: Dynamic PET/CT Imaging

INTERVENTIONS:
Device: Dynamic PET/CT Imaging — -Will take approximately 60 minutes

SUMMARY:
The goal of this study is to see how the images collected during the first hour compare with the routine images collected as part of the clinical scan.

ELIGIBILITY:
Inclusion Criteria Main Cohort:

* 18 years of age or older
* Scheduled to undergo a clinical PET/CT scan with any clinically prescribed radiotracer for known or suspected malignancy (pathologic confirmation not required)
* Able to provide informed consent

Inclusion Criteria Repeatability Cohort:

* 18 years of age or older
* Scheduled to undergo a clinical PET/CT FDG or 68Ga- DOTA-0-Tyr3-Octreotate (DOTATATE) for known or suspected malignancy (pathologic confirmation not required)
* Able to provide informed consent

Exclusion Criteria:

-Younger than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-05-29 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Wahl, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators may share your images with other researchers. They may be doing research in areas similar to this research or in other unrelated areas. These researchers may be at Washington University, at other research centers and institutions, or industry sponsors of research. The investigators may also share your research data with large data repositories (a repository is a database of information) for broad sharing with the research community. If the individual research data is placed in one of these repositories only qualified researchers, who have received prior approval from individuals that monitor the use of the data, will be able to look at the information.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Beginning 3 months and ending 10 years following article publication.
Access Criteria: Proposals should be directly submitted to rwahl@wustl.edu.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dynamic PET Imaging
Started | 80
Completed | 80
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Dynamic PET Imaging
Number analyzed (Participants) | 80
Age, Continuous [Median (Full Range); unit: years] | 66 [33 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 78
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 75
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 80

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Rapid, Whole-body Dynamic PET Imaging as Measured by Number of Participants Who Successfully Completed the Study Imaging Component
Description: -Successful completion of the study imaging component will be defined as: (1) patient remains on scanner for the full dynamic phase of PET imaging prior to the standard of care PET/CT and (2) automated scanner software is able to successfully generate valid parametric maps (requires at least three consecutive whole-body PET acquisitions without substantial motion between acquisitions).
Time Frame: At time of scan (day 1)
Measure: Count of Participants; unit: Participants
Arm/Group | Dynamic PET Imaging
Number analyzed (Participants) | 80
Participants | 80

2. Secondary Outcome: Quantitative Impacts of Data Motion Correction (OncoFreeze) as Measured by Semi-quantitative Standardized Uptake Value (SUV)-Max
Description: Subjects underwent standard-of-care (SOC) PET acquisition with a respiratory-gating belt. Ungated (UG), belt-gating-derived optimal gate (BG-OG), EMCD utilizing belt gating (BG-EMCD), and EMCD utilizing data-driven gating (DDG-EMCD) images were reconstructed. Tracer-avid lesions in the lower chest or upper abdomen were segmented. Quantitative metrics were extracted.
Time Frame: At the time of scan (Day 1)
Population: This outcome measure requires subjects to have disease so only 36 subjects had disease.
Measure: Median (Inter-Quartile Range); unit: SUV-max
Arm/Group | Dynamic PET Imaging
Number analyzed (Participants) | 36
SUV-max
  Belt-gating optimal gate | 10.77 [6.21 to 18.46]
  Elastic motion correction with blurring utilizing belt gating | 10.75 [5.86 to 18.70]
  Elastic motion correction with blurring utilizing data-driven gating | 10.74 [6.04 to 18.66]
  Ungated | 9.00 [5.01 to 15.97]

3. Secondary Outcome: Quantitative Impacts of Data Motion Correction (OncoFreeze) as Measured by Lesion Contrast-to-noise Ratios (CNRs)
Description: as for outcome 2
Time Frame: At the time of scan (Day 1)
Population: This outcome measure required subjects to have cancer so only 36 subjects had sufficient cancer in order to be analyzed.
Measure: Median (Inter-Quartile Range); unit: contrast-to-noise ratio
Arm/Group | Dynamic PET Imaging
Number analyzed (Participants) | 36
contrast-to-noise ratio
  Belt-gating optimal gate | 6.31 [3.97 to 12.08]
  Elastic motion correction with blurring utilizing belt gating | 9.14 [5.59 to 15.87]
  Elastic motion correction with blurring utilizing data-driven gating | 8.89 [5.50 to 17.05]
  Ungated | 7.89 [4.99 to 15.17]

4. Secondary Outcome: Clinical Impacts of Data Motion Correction (OncoFreeze) as Measured by Mean Relative Lesion Number Between Ungated and Belt-gating Optimal Gate
Description: * Will be assessed by Reader 1 and Reader 2 by comparing motion-corrected images derived from OncoFreeze with standard static non-gated PET images and conventionally gated PET images.
  * OncoFreeze is a novel approach to PET motion correction that utilizes 100% of events, which are corrected to an optimal gate image utilizing an optical flow algorithm, creating the potential for motion corrected images without increasing image noise.
Time Frame: At the time of scan (Day 1)
Population: This outcome measure required subjects to have cancer so only 36 subjects had sufficient cancer in order to be analyzed.
Measure: Mean (Full Range); unit: relative lesions
Groups:
- Dynamic PET Imaging Ungated; Dynamic PET/CT Belt-Gating Optimal Gate: * Dynamic PET/CT imaging will begin at approximately the same time as the clinically prescribed radiotracer injection and will continue until approximately the start of the clinical scan
  * A subset of patients (up to 30 scheduled to undergo FDG or DOTATATE PET/CT imaging) will be asked to return within 7 days for a repeat imaging study.
Arm/Group | Dynamic PET Imaging Ungated | Dynamic PET/CT Belt-Gating Optimal Gate
Number analyzed (Participants) | 36 | 36
relative lesions
  Reader 1 | 1.11 [0 to 9] | 0.14 [0 to 9]
  Reader 2 | 0.31 [0 to 2] | 0.14 [0 to 2]
Statistical Analysis 1: Comparison: Dynamic PET Imaging Ungated vs Dynamic PET/CT Belt-Gating Optimal Gate; This statistical analysis is for Reader 1; Test type: Superiority; p = 0.001, Two-tailed Wildoxon signed-rank test
Statistical Analysis 2: Comparison: Dynamic PET Imaging Ungated vs Dynamic PET/CT Belt-Gating Optimal Gate; This statistical analysis is for Reader 2; Test type: Superiority; p = 0.28, Two-tailed Wilcoxon signed-rank test

5. Secondary Outcome: Clinical Impacts of Data Motion Correction (OncoFreeze) as Measured by Mean Relative Lesion Number Between Ungated and Elastic Motion Correction With Blurring Utilizing Belt Gating
Description: as for outcome 4
Time Frame: At the time of scan (Day 1)
Population: This outcome measure required subjects to have cancer so only 36 subjects had sufficient cancer in order to be analyzed.
Measure: Mean (Full Range); unit: mean relative lesion number
Groups:
- Dynamic PET/CT Elastic Motion Correction With Blurring Utilizing Belt Gating: * Dynamic PET/CT imaging will begin at approximately the same time as the clinically prescribed radiotracer injection and will continue until approximately the start of the clinical scan
  * A subset of patients (up to 30 scheduled to undergo FDG or DOTATATE PET/CT imaging) will be asked to return within 7 days for a repeat imaging study.
Arm/Group | Dynamic PET Imaging Ungated | Dynamic PET/CT Elastic Motion Correction With Blurring Utilizing Belt Gating
Number analyzed (Participants) | 36 | 36
mean relative lesion number
  Reader 1 | 1.11 [0 to 9] | 1.28 [0 to 9]
  Reader 2 | 0.31 [0 to 2] | 0.50 [0 to 2]
Statistical Analysis 1: Comparison: Dynamic PET Imaging Ungated vs Dynamic PET/CT Elastic Motion Correction With Blurring Utilizing Belt Gating; This is the statistical analysis for Reader 1; Test type: Superiority; p = 0.22, Two-tailed Wilcoxon signed-rank test
Statistical Analysis 2: Comparison: Dynamic PET Imaging Ungated vs Dynamic PET/CT Elastic Motion Correction With Blurring Utilizing Belt Gating; This is the statistical analysis for Reader 2; Test type: Superiority; p > 0.05, Two-tailed Wilcoxon signed-rank test

6. Secondary Outcome: Clinical Impacts of Data Motion Correction (OncoFreeze) as Measured by Mean Relative Lesion Number Between Ungated and Elastic Motion Correction With Blurring Utilizing Data-driven Gating
Description: as for outcome 4
Time Frame: At the time of scan (Day 1)
Population: This outcome measure required subjects to have cancer so only 36 subjects had sufficient cancer in order to be analyzed.
Measure: Mean (Full Range); unit: mean relative lesion number
Groups:
- Dynamic PET/CT Elastic Motion Correction With Blurring Utilizing Data-Driven Gating: * Dynamic PET/CT imaging will begin at approximately the same time as the clinically prescribed radiotracer injection and will continue until approximately the start of the clinical scan
  * A subset of patients (up to 30 scheduled to undergo FDG or DOTATATE PET/CT imaging) will be asked to return within 7 days for a repeat imaging study.
Arm/Group | Dynamic PET Imaging Ungated | Dynamic PET/CT Elastic Motion Correction With Blurring Utilizing Data-Driven Gating
Number analyzed (Participants) | 36 | 36
mean relative lesion number
  Reader 1 | 1.11 [0 to 9] | 1.47 [0 to 9]
  Reader 2 | 0.31 [0 to 2] | 0.50 [0 to 2]
Statistical Analysis 1: Comparison: Dynamic PET Imaging Ungated vs Dynamic PET/CT Elastic Motion Correction With Blurring Utilizing Data-Driven Gating; This is the statistical analysis for Reader 1; Test type: Superiority; p = 0.009, Two-tailed Wilcoxon signed-rank test
Statistical Analysis 2: Comparison: Dynamic PET Imaging Ungated vs Dynamic PET/CT Elastic Motion Correction With Blurring Utilizing Data-Driven Gating; This statistical analysis is for Reader 2; Test type: Superiority; p > 0.05, Two-tailed Wilcoxon signed-rank test

7. Secondary Outcome: Clinical Impacts of Data Motion Correction (OncoFreeze) as Measured by Mean Relative Lesion Number Between Belt-gating Optimal Gate and Elastic Motion Correction With Blurring Utilizing Belt Gating
Description: * Will be assessed by Reader 1 and Reader 2 comparing motion-corrected images derived from OncoFreeze with standard static non-gated PET images and conventionally gated PET images.
  * OncoFreeze is a novel approach to PET motion correction that utilizes 100% of events, which are corrected to an optimal gate image utilizing an optical flow algorithm, creating the potential for motion corrected images without increasing image noise.
Time Frame: At the time of scan (Day 1)
Population: This outcome measure required subjects to have cancer so only 36 subjects had sufficient cancer in order to be analyzed.
Measure: Mean (Full Range); unit: mean relative lesion number
Groups:
- Dynamic PET Imaging Belt-gating Optimal Gate; Dynamic PET/CT Elastic Motion Correction With Blurring Utilizing Belt Gating: * Dynamic PET/CT imaging will begin at approximately the same time as the clinically prescribed radiotracer injection and will continue until approximately the start of the clinical scan
  * A subset of patients (up to 30 scheduled to undergo FDG or DOTATATE PET/CT imaging) will be asked to return within 7 days for a repeat imaging study.
Arm/Group | Dynamic PET Imaging Belt-gating Optimal Gate | Dynamic PET/CT Elastic Motion Correction With Blurring Utilizing Belt Gating
Number analyzed (Participants) | 36 | 36
mean relative lesion number
  Reader 1 | 0.14 [0 to 1] | 1.28 [0 to 9]
  Reader 2 | 0.14 [0 to 2] | 0.50 [0 to 2]
Statistical Analysis 1: Comparison: Dynamic PET Imaging Belt-gating Optimal Gate vs Dynamic PET/CT Elastic Motion Correction With Blurring Utilizing Belt Gating; This is the statistical analysis for Reader 1; Test type: Superiority; p < 0.001, Two-tailed Wilcoxon signed-rank test
Statistical Analysis 2: Comparison: Dynamic PET Imaging Belt-gating Optimal Gate vs Dynamic PET/CT Elastic Motion Correction With Blurring Utilizing Belt Gating; This is the statistical analysis for Reader 2; Test type: Superiority; p = 0.02, Two-tailed Wilcoxon signed-rank test

8. Secondary Outcome: Clinical Impacts of Data Motion Correction (OncoFreeze) as Measured by Mean Relative Lesion Number Between Belt-gating Optimal Gate and Elastic Motion Correction With Blurring Utilizing Data-driven Gating
Description: * Will be assessed Reader 1 and Reader 2 by comparing motion-corrected images derived from OncoFreeze with standard static non-gated PET images and conventionally gated PET images.
  * OncoFreeze is a novel approach to PET motion correction that utilizes 100% of events, which are corrected to an optimal gate image utilizing an optical flow algorithm, creating the potential for motion corrected images without increasing image noise.
Time Frame: At the time of scan (Day 1)
Population: This outcome measure required subjects to have cancer so only 36 subjects had sufficient cancer in order to be analyzed.
Measure: Mean (Full Range); unit: mean relative lesion number
Arm/Group | Dynamic PET Imaging Belt-gating Optimal Gate | Dynamic PET/CT Elastic Motion Correction With Blurring Utilizing Data-driven Gating
Number analyzed (Participants) | 36 | 36
mean relative lesion number
  Reader 1 | 0.14 [0 to 1] | 1.47 [0 to 9]
  Reader 2 | 0.14 [0 to 2] | 0.50 [0 to 2]
Statistical Analysis 1: Comparison: Dynamic PET Imaging Belt-gating Optimal Gate vs Dynamic PET/CT Elastic Motion Correction With Blurring Utilizing Data-driven Gating; This is the statistical analysis for Reader 1; Test type: Superiority; p < 0.001, Two-tailed Wilcoxon signed-rank test
Statistical Analysis 2: Comparison: Dynamic PET Imaging Belt-gating Optimal Gate vs Dynamic PET/CT Elastic Motion Correction With Blurring Utilizing Data-driven Gating; This is the statistical analysis for Reader 2; Test type: Superiority; p = 0.02, Two-tailed Wilcoxon signed-rank test

9. Secondary Outcome: Clinical Impacts of Data Motion Correction (OncoFreeze) as Measured by Mean Relative Lesion Number Between Elastic Motion Correction With Blurring Utilizing Belt Gating and Elastic Motion Correction With Blurring Utilizing Data-driven Gating
Description: as for outcome 4
Time Frame: At the time of scan (Day 1)
Population: This outcome measure required subjects to have cancer so only 36 subjects had sufficient cancer in order to be analyzed.
Measure: Mean (Full Range); unit: mean relative lesion number
Groups:
- Dynamic PET Imaging Elastic Motion Correction With Blurring Utilizing Belt Gating; Dynamic PET/CT Elastic Motion Correction With Blurring Utilizing Data-driven Gating: * Dynamic PET/CT imaging will begin at approximately the same time as the clinically prescribed radiotracer injection and will continue until approximately the start of the clinical scan
  * A subset of patients (up to 30 scheduled to undergo FDG or DOTATATE PET/CT imaging) will be asked to return within 7 days for a repeat imaging study.
Arm/Group | Dynamic PET Imaging Elastic Motion Correction With Blurring Utilizing Belt Gating | Dynamic PET/CT Elastic Motion Correction With Blurring Utilizing Data-driven Gating
Number analyzed (Participants) | 36 | 36
mean relative lesion number
  Reader 1 | 1.28 [0 to 9] | 1.47 [0 to 9]
  Reader 2 | 0.50 [0 to 2] | 1.47 [0 to 9]

10. Secondary Outcome: Repeatability of Dynamic Imaging as Measured by Calculating the Measurement Agreement in Semi-quantitative PET Metrics Between Test and Retest Dynamic Images
Description: * Standardized uptake value (SUV)-max, SUV-peak, Uptake time-corrected SUV (cSUV), Standardized uptake ratio (SUR), Uptake time-corrected standardized uptake ratio (cSUR), Patlak slope (PS)-max, and PS-peak were analyzed.
  * Test-retest repeatability of quantitative metrics based on the PS versus the SUV among lesions and normal organs on oncologic [18F]FDG-PET/CT.
  * Repeatability was assessed via mean test-retest percent changes [T-RT %Δ]
Time Frame: Day 1 and approximately 1 week later
Population: Only 9 subjects completed the test-retest protocol and of those only 4 subjects had [18F]FDG-avid lesions.
Measure: Mean (95% Confidence Interval); unit: test-retest percent changes
Arm/Group | Dynamic PET Imaging
Number analyzed (Participants) | 4
test-retest percent changes
  PS-max | 11 [-32 to 54]
  PS-peak | 15 [-30 to 59]
  SUV-max | 47 [3 to 91]
  SUV-peak | 26 [-22 to 75]
  cSUV-max | -6 [-53 to 41]
  cSUV-peak | -27 [-77 to 23]
  SUR-max | 81 [48 to 114]
  SUR-peak | 63 [23 to 102]
  cSUR-max | 7 [-33 to 48]
  cSUR-peak | -14 [-60 to 33]

11. Secondary Outcome: Metabolic Rate of Images
Description: -Will help to determine the optimal post-injection time period for dynamic PET imaging for Early (35-50 min post-injection) and Late (75-90 min post-injection) Patlak slope (PS) analysis. Reader 1 and Reader 2 used a standard Likert score from 0-4 with 1 being the worst and 4 being the best. A higher score indicated the image was easier to read.
Time Frame: At the time of scan (Day 1)
Population: This outcome measure required subjects to have cancer so only 41 subjects had sufficient cancer in order to be analyzed.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Dynamic PET Imaging
Number analyzed (Participants) | 41
score on a scale
  PS-Early Reader 1 | 1.19 [1 to 2]
  PS-Late Reader 1 | 3.95 [3 to 4]
  PS-Early Reader 2 | 2.14 [1 to 4]
  PS-Late Reader 2 | 3.95 [3 to 4]
Statistical Analysis 1: Comparison: Dynamic PET Imaging; This is the statistical analysis comparing PS-Early Reader 1 to PS-Late Reader 1; Test type: Superiority; p < 0.001, Two-tailed Wilcoxon signed-rank test
Statistical Analysis 2: Comparison: Dynamic PET Imaging; This is the statistical analysis comparing PS-Early Reader 2 and PS-Late Reader 2; Test type: Superiority; p < 0.001, Two-tailed Wilcoxon signed-rank test

12. Secondary Outcome: Volume of Distribution (Intercept) Images
Description: -Will help to determine the optimal post-injection time period for dynamic PET imaging for Patlak analysis.
Time Frame: At the time of scan (Day 1)
Population: The intercept images were unacceptable due to high quantitative biases and noise levels.
Arm/Group | Dynamic PET Imaging
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events and all-cause mortality were collected on the day of the PET/CT.
Arm/Group | Dynamic PET Imaging
All-Cause Mortality (participants affected / at risk) | 0/80
Serious Adverse Events (participants affected / at risk) | 0/80
Other Adverse Events (participants affected / at risk) | 1/80
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dynamic PET Imaging (N=80)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-20): https://cdn.clinicaltrials.gov/large-docs/52/NCT04283552/Prot_SAP_000.pdf